CLINICAL TRIAL: NCT01861457
Title: Reduction of Staph Aureus Carriage by Non-Antibiotic NOZIN® Nasal Sanitizer®
Brief Title: Reduction of Staph Aureus Carriage by Non-Antibiotic NOZIN® Nasal Sanitizer® Antiseptic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Shaun A. Nguyen, MD, Associate Professor- Department of Otolaryngology - Head and Neck Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nozin
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Infectious Disease
Keywords: nasal sanitizer®; S. aureus; general bacteria; nasal carriage; decolonization
MeSH Terms: conditions — Communicable Diseases; Staphylococcal Infections | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nozin® Nasal Sanitizer® (Experimental): Non-antibiotic, alcohol-based antiseptic
  Interventions: Other: Nozin® Nasal Sanitizer®
- Phosphate-buffered saline (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Nozin® Nasal Sanitizer® — The treatment agent tested was the alcohol and natural oil preparation that comprises the commercially available over-the-counter (OTC) product, NOZIN® Nasal Sanitizer® antiseptic, by Global Life Technologies Corp, with the addition of benzalkonium chloride (0.13%), as described for the patented and safety-tested formulation.
  Other Names: Nozin® Nasal Sanitizer® antiseptic
  Arms: Nozin® Nasal Sanitizer®
Other: Placebo — The placebo preparation, utilized to account for the potential mechanical effects of the application process, was phosphate buffered saline (PBS).
  Other Names: Sham
  Arms: Phosphate-buffered saline

SUMMARY:
The purpose of this study is to determine the extent to which bacterial growth in the nostrils by S. aureus, a common bacteria that is found in hospital environment, can be reduced by NOZIN® Nasal Sanitizer® antiseptic nasal swabs during the course of a typical 10-hour work period in participants known to have S. aureus in their nose passages.

DETAILED DESCRIPTION:
The purpose of the proposed pilot study is to employ a repeated sampling protocol to test the effectiveness of a currently marketed, over-the-counter topical preparation to reduce carriage of Staphylococcus aureus (S. aureus) in the nasal vestibules of health professionals working in an outpatient clinical setting. The product to be tested is the NOZIN® Nasal Sanitizer® antiseptic produced by Global Life Technologies Corp. It is an alcohol-based, non-antibiotic antiseptic preparationl

The study has one primary Specific Aim:

To determine the extent to which colonization of the vestibular region of the nares by S. aureus can be reduced by a regimen of nasal topical applications of the alcohol-based antiseptic during the course of typical 10-hour work day in subjects known to exhibit S. aureus nasal carriage.

A secondary aim of the study will be to evaluate the concurrent effectiveness of the antiseptic applications on a measure of general bacterial colonization within the vestibules of each subject.

ELIGIBILITY:
Inclusion Criteria:

* All healthy health care professionals between the ages of 18 and 60 years of age who are regular full-time employees of the MUSC Hospital, work a 10 or 12 hour work shift, and test positive for nasal vestibular S. aureus carriage within 10 days prior to their scheduled study day will be eligible to participate in the study.

Exclusion Criteria:

* Excluded from the study will be individuals exhibiting symptoms of upper respiratory disease, including chronic rhinitis/sinusitis, seasonal allergies, upper respiratory infection during the previous four weeks, have known allergy to citrus or soy oil, or are "smokers". "Non-smokers" will be defined as those individuals who have abstained from smoking for at least one year prior to the study. Subjects must be able and agree to refrain from using prescription and non-prescription nasal spray or other nasal preparations or washes from the time of their screening up to and during their scheduled study day.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun A Nguyen, MD, Principal Investigator — Medical University of South Carolina- Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Steed LL, Costello J, Lohia S, Jones T, Spannhake EW, Nguyen S. Reduction of nasal Staphylococcus aureus carriage in health care professionals by treatment with a nonantibiotic, alcohol-based nasal antiseptic. Am J Infect Control. 2014 Aug;42(8):841-6. doi: 10.1016/j.ajic.2014.04.008. Epub 2014 Jun 2. PMID 24881497
- See also: Site containing information regarding the alcohol-based antiseptic preparation used — http://www.nozin.com
- See also: Site containing information regarding the alcohol-based antiseptic preparation used — http://www.nozinpro.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants came from the nursing and technical staff working in the Main and Ambulatory operating rooms and patient care floors of the MUSC Hospital. Eligible to participate in the study were all healthy individuals between the ages of 18 and 70 years of age who were regular full-time employees working a minimum 10-hour workday.
Pre-assignment Details: Following the initial interview and after obtaining informed written consent, eligible subjects were screened to identify those who demonstrated nasal vestibular carriage of S. aureus. Subjects testing positive were invited to enroll in the study protocol within the subsequent 10 days.
Groups:
- Nozin® Nasal Sanitizer®: Participants undergo three nasal vestibular applications of the alcohol-based antiseptic using a saturated nasal swab at 4-hour intervals during the 10-hour study period.
- Phosphate-buffered Saline (PBS) Placebo: Participants undergo three nasal vestibular applications of the PBS placebo using a saturated nasal swab at 4-hour intervals during the 10-hour study period.
Period: Overall Study
Arm/Group | Nozin® Nasal Sanitizer® | Phosphate-buffered Saline (PBS) Placebo
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nozin Nasal Sanitizer: Apply 4 rotations of swab to each nostril 3x in a 10-hour study period.
  Nozin Nasal Sanitizer
- Saline Placebo: Apply 4 rotations of swab to each nostril 3x in a 10-hour study period.
  Placebo
- Total: Total of all reporting groups
Arm/Group | Nozin Nasal Sanitizer | Saline Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Full Range); unit: years] | 34.5 [26 to 64] | 35.4 [26 to 67] | 35.1 [26 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Treatment-associated Change in S. Aureus Colonization During a Typical 10-hour Work Day
Description: The percent change from morning baseline sample to the evening sample taken at the end of a typical 10-hour workday in treated subjects known to be colonized by Staph aureus.
Time Frame: 10-hour work day
Population: All participants who received 3 scheduled treatments
Measure: Median (Inter-Quartile Range); unit: Percent change in colonization
Groups:
- Alcohol-Based Nasal Antiseptic: Participants known to exhibit Staph aureus carriage by previous nasal swab screening and randomly assigned received application by nasal swab of alcohol-based nasal antiseptic (Nozin® Nasal Sanitizer®) at 0, 4 and 8 hrs.
- Placebo: Participants known to exhibit Staph aureus carriage by previous nasal swab screening and randomly assigned received application of placebo treatment with phosphate-buffered saline at 0, 4 and 8 hrs.
Arm/Group | Alcohol-Based Nasal Antiseptic | Placebo
Number analyzed (Participants) | 20 | 19
Percent change in colonization | -99.8 [-100 to -80.6] | -13.5 [-69.3 to 149.4]
Statistical Analysis 1: Comparison: Alcohol-Based Nasal Antiseptic vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Treatment-associated Change in Total Nasal Bacterial Colonization During a Typical 10-hour Work Day
Description: as for outcome 1
Time Frame: 10 hour workday
Measure: Median (Inter-Quartile Range); unit: Percent change in colonization
Arm/Group | Alcohol-Based Nasal Antiseptic | Placebo
Number analyzed (Participants) | 20 | 19
Percent change in colonization | -91.0 [-97.2 to -72.0] | 24.0 [-63.4 to 74.6]
Statistical Analysis 1: Comparison: Alcohol-Based Nasal Antiseptic vs Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Over the 10 hour period of applications
Description: Serious: allergic symptoms; Other: nasal dryness, irritation, burning.
Groups:
- Nozin Nasal Sanitizer: Apply 4 rotations of swab to each nostril every four hours
  Nozin Nasal Sanitizer
- Sham: Apply 4 rotations of swab to each nostril every four hours ...
  Sham
Arm/Group | Nozin Nasal Sanitizer | Sham
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No